CLINICAL TRIAL: NCT00585611
Title: Effects of Statin Therapy on Vascular Properties and Outcomes in Diastolic Heart Failure Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit into the study
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2005-0430
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Diastolic Heart Failure
Keywords: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): Heart failure patients assigned to atorvastatin
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: Atorvastatin; Other: placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin - 40 mg orally daily for 6 months
Other: placebo — placebo
  Arms: 2

SUMMARY:
The study is designed to define the underlying vascular abnormalities present in patients with diastolic heart failure and test the effect of a therapy aimed at vascular abnormalities. This study is designed to investigate the effects of therapy with atorvastatin in subjects with diastolic heart failure to improve abnormalities of vascular and myocardial structure and function, with particular emphasis on arterial stiffness and endothelial dysfunction.

DETAILED DESCRIPTION:
Forty subjects will be given either drug (atorvastatin 40 mg) or placebo in a randomized fashion once daily for six months. Using echocardiography, tonometry, and flow mediated dilation of conduit arteries and arterioles, baseline cardiovascular anatomy and physiology will be defined. Subjects that enroll in the study will be required to come in for 5 study visits. The initial visit is a screening visit; subject consent is obtained and an echocardiogram is performed as well as blood tests. At the randomization visit (4-14 days following screening), the subject will be provided with drug or placebo in a blinded fashion.Also at this visit, subjects will be asked to do a 6 minute walk, QOL questionnaire, and vascular function testing. There will be follow-up study visits at 1 and 3 months following randomization. At each follow-up visit a medical history, pill count and brief physical examination will be performed, a repeat QOL questionnaire administered, and blood tests to assess safety of the statin therapy. At 6 months, the final study visit will occur. At this visit a full history and detailed physical examination will be performed. Repeat echocardiogram, 6 minute walk test, QOL questionnaire, and vascular function examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Age > 18,
* Ejection fraction ≥ 50%,
* hospitalization for heart failure in the last 6 months and
* current NYHA Class II-IV symptoms, OR
* current NYHA Class III-IV symptoms and one of the following:

  1. ECG or echocardiographic evidence of moderate/severe left ventricular hypertrophy,
  2. chest x-ray evidence of pulmonary congestion

Exclusion Criteria:

* Probable alternative cause of symptoms (pulmonary disease, severe anemia, etc.)
* Prior documented LVEF < 40% or qualitative moderate or greater LV systolic dysfunction.
* Current indication for statin therapy
* Intolerance to statin therapy.
* Documented ischemic heart disease requiring lipid-lowering therapy (i.e. CAD, myocardial infarction, stroke)
* Evidence of significant myocardial ischemia on stress testing at screening visit.
* Evidence of hepatic abnormality (defined as liver enzymes > 2 times the upper limit of normal values).
* Uncontrolled hypertension (BP > 150/100)
* Significant valvular disease.
* Atrial fibrillation
* Known familial hypertrophic cardiomyopathy or obstructive hypertrophic cardiomyopathy.
* Restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease (i.e. amyloidosis, sarcoidosis, hemochromatosis).
* Cor pulmonale or other cause of right heart failure not related to LV dysfunction.
* Clinically significant pulmonary disease.
* Pericardial constriction or hemodynamically significant pleural effusion.
* Uncontrolled arrhythmia.
* Any systemic condition other than heart failure that may limit survival to less than 2 years.
* Advance renal disease (serum creatinine > 3.0 mg/dl or on dialysis)
* Known intolerance or allergy to HMG CoA reductase inhibitors
* Uncontrolled hyper- or hypothyroidism.
* Any subject characteristic that may interfere with study compliance, such as baseline dementia, substance abuse, history of non-compliance with medications or appointments.
* Prisoners or other vulnerable populations.
* Any woman of child-bearing age with a documented positive pregnancy test.
* Subject is receiving therapy with other investigational therapy or is participating in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the record documents 1 participant enrolled in this study, there are no data available to report.
Groups:
- Arm 2: Atorvastatin: Atorvastatin - 40 mg orally daily for 6 months
  placebo: placebo
Period: Overall Study
Arm/Group | Atorvastatin | Arm 2
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There are no data available
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Arm 2 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotid-femoral Pulse Wave Velocity (CFPWV) in the Statin Treated vs. Control Group
Time Frame: 6 months after initiation of intervention
Population: There are no data available
Arm/Group | Atorvastatin | Arm 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Composite Cardiovascular Endpoint Incorporating Quality of Life (QOL) Assessment + Hospitalizations for Cardiovascular Disease and Mortality
Time Frame: 6 months after initiation of intervention
Population: There are no data available.
Arm/Group | Atorvastatin | Arm 2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Changes in Submaximal Exercise Capacity Measured by 6-minute Walk Test
Time Frame: 6 months after initiation of intervention
Population: There are no data available.
Arm/Group | Atorvastatin | Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: There are no data available
Description: There are no data available to report.
Arm/Group | Atorvastatin | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
PI left UW-Madison, has no data for participant enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes